CLINICAL TRIAL: NCT00606281
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group-Comparison Trial of Aripiprazole in the Treatment of Patients With Bipolar Disorder Experiencing a Manic or Mixed Episode
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 031-06-003
Record Dates: First submitted 2008-01-19; First posted 2008-02-01 (Estimated); Results first posted 2014-02-12 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-01

CONDITIONS: Bipolar I Disorder
MeSH Terms: interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Aripiprazole
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Aripiprazole — oral, 24mg/day
  Other Names: OPC-14597
  Arms: 1
Drug: placebo — oral, 0mg(4tablets)/day
  Other Names: OPC-14597
  Arms: 2

SUMMARY:
The primary objective of this trial is to evaluate the clinical efficacy and safety of aripiprazole in comparison to placebo in patients with Bipolar I Disorder experiencing a manic or mixed episode.

ELIGIBILITY:
Inclusion Criteria:

* Trial subjects will be men and women of age 18 or above and below the age of 65 who will not be turning 65 during the trial.
* Patients have the ability to understand and to provide informed consent to the examination, observation, and evaluation processes specified in this protocol, and have signed the informed consent form based on a full understanding of the trial.
* Patients who meet DSM-IV-TR criteria for manic or mixed episodes and have been diagnosed as having "296.4x Bipolar I Disorder in which the most recent episode was manic" or "296.6x Bipolar I Disorder in which the most recent episode was mixed"
* Patients with a YMRS total score of 20 or more

Exclusion Criteria:

* Patients presenting with a clinical picture and/or history that is consistent with a DSM-IV-TR diagnosis of:

  * Delirium, dementia, amnestic disorder, or other cognitive disorders
  * Schizophrenia or other psychotic disorder
  * Personality disorder
* Patients experiencing their first manic or mixed episode
* Patients whose current manic episode has lasted for more than 4 weeks
* Patients with psychotic symptoms that are clearly due to another general medical condition or direct physiological effects of a substance
* Patients who have met DSM-IV-TR criteria for a substance-related disorder within 3 months (90 days) prior to informed consent (excluding caffeine- and nicotine-related disorders, but including abuse of benzodiazepines)
* Patients who have received ECT treatment within 8 weeks prior to informed consent
* Patients who are expected to require administration of ultrashort-acting or short-acting benzodiazepine receptor agonist hypnotics and antianxiety drugs (See (1) of 4.2.2) at doses exceeding the equivalent of 15 mg/day of diazepam (Only for those patients using such drugs)
* Patients at significant risk of developing a severe adverse event. Patients who have a medical condition that would interfere with assessments of safety or efficacy during the course of the trial, or who have a history of such a condition.
* Patients who have received any of the following treatments during the screening period:

  * Reserpine
  * Levodopa, dopamine receptor stimulants
  * Monoamine oxidase inhibitors
  * Psychostimulants
  * Thyroid hormones, antithyroid drugs
  * Corticosteroids (other than topical preparations)
  * Adrenaline
  * All other investigational or unapproved agents
  * ECT
  * Light therapy
* For patients who take lithium, valproate, or carbamazepine within 3 days prior to commencement of investigational product administration, those patients with serum concentrations of lithium greater than 0.6 mmol/L, serum concentrations of valproate greater than 50 µg/mL, or serum concentrations of carbamazepine greater than 4 µg/mL
* Patients judged to have a diabetic blood glucose level (judgment based on use of a self-monitoring blood glucose meter permissible), or patients whose HbA1c is 6.5% or higher
* Patients with a history or a complication of diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2008-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Saito, Study Director — Department of Clinical Research and Development, Division of New Product Evaluation and Development
Locations (12):
- Hong Kong, China
- Japan (9):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Hokuriku Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region
- Seoul, South Korea
- Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Groups:
- Aripiprazole: Subjects were administered 24 mg/day of aripiprazole once daily for 21 days. If there was a problem with tolerability, the dose could be reduced to 12 mg/day.
- Placebo: Subjects were administered placebo once daily for 21 days.
Period: Overall Study
Arm/Group | Aripiprazole | Placebo
Started | 128 | 130
Completed | 72 | 64
Not Completed | 56 | 66
Not completed — Adverse Event | 11 | 12
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 28 | 35
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 3 | 3
Not completed — Withdrawal by Subject | 11 | 13
Not completed — Progression to depressive phase | 1 | 1
Not completed — Change of residence or other commitments | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Population(FAS)：
  Excluding the following subjects from the randomized subjects:
  * 2 subjects who did not take the study medication (Aripipirazole:1, Placebo:1)
  * 8 subjects with GCP violation (Aripipirazole:5, Placebo:3)
  * 1 subject whose post dose efficacy were not available (Placebo:1)
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole | Placebo | Total
Number analyzed (Participants) | 122 | 125 | 247
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (12.46) | 37.8 (12.69) | 37.6 (12.50)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 2 | 5
  Between 18 and 65 years | 119 | 123 | 242
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 75 | 145
  Male | 52 | 50 | 102
Region of Enrollment [Number; unit: participants]
  Taiwan | 17 | 18 | 35
  China | 28 | 28 | 56
  Japan | 39 | 40 | 79
  Indonesia | 7 | 8 | 15
  Malaysia | 12 | 13 | 25
  Philippines | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Young Mania Rating Scale (YMRS)
Description: Using LOCF datasets, change in YMRS total score from baseline (Day 1) to endpoint (Day 21) was evaluated through analysis of covariance(ANCOVA).
  YMRS is composed of 11 evaluation items with 5 rating levels each. Items rated on a scale of 0 to 4 (comprising 5 rating levels of one point each) are 1) elevated mood, 2) increased motor activity/energy, 3) sexual interest, 4) sleep, 7) language-thought disorder, 10) appearance, and 11) insight. Items rated on a scale of 0 to 8 (comprising 5 rating levels of two points each) are 5) irritability, 6) speech (rate and amount), 8) content, and 9) disruptive-aggressive behavior.
  YMRS ranges from 0 (best possible outcome) to 60 (worst possible outcome).
Time Frame: Day1, Day21
Population: Full analysis set (FAS): The FAS consisted of subjects who had received at least one dose of investigational product and for whom the post-dosing efficacy parameter data had been obtained. Cases of GCP violation were excluded from analysis.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 122 | 125
scores on a scale | -11.3 (1.31) | -5.3 (1.29)
Statistical Analysis 1: Comparison: Aripiprazole vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -6.0, 95% CI 2-sided [-9.4 to -2.7]

2. Secondary Outcome: Clinical Global Impression - Bipolar Version (CGI-BP), Severity of Illness Score (Mania)
Description: CGI-BP severity of illness is a scale for overall evaluation of the severity of bipolar disorder; it comprises 3 components-mania, depression, and overall bipolar illness.
  CGI-BP severity of illness score (mania) ranges form 1 (normal, not ill) to 7 (very severely ill).
  Using LOCF datasets, change in CGI-BP severity of illness score (mania) from baseline (Day 1) to endpoint (Day 21) was evaluated through ANCOVA.
Time Frame: Day1, Day21
Population: FAS: The FAS consisted of subjects who had received at least one dose of investigational product and for whom the post-dosing efficacy parameter data had been obtained. Cases of GCP violation were excluded from analysis.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 122 | 125
scores on a scale | -1.4 (0.15) | -0.7 (0.15)
Statistical Analysis 1: Comparison: Aripiprazole vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.7, 95% CI [-1.1 to -0.3]

ADVERSE EVENTS:
Time Frame: 21 weeks
Description: 1 subject in the placebo group took the study medication (aripiprazole) before proper randomization and was later assigned to the placebo group by IVRS. It was decided to include this subject in the aripiprazole group for safety analysis. However, she was included in the placebo group for the FAS.
Arm/Group | Aripiprazole | Placebo
Serious Adverse Events (participants affected / at risk) | 5/123 | 9/125
Other Adverse Events (participants affected / at risk) | 69/123 | 45/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole (N=123) | Placebo (N=125)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Multiple Fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bipolar Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Bipolar I Disorder (Psychiatric disorders) | 1 (1) | 4 (4)
Mania (Psychiatric disorders) | 3 (3) | 4 (4)
Drug Erption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole (N=123) | Placebo (N=125)
Constipation (Gastrointestinal disorders) | 10 (11) | 8 (9)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 7 (8)
Nausea (Gastrointestinal disorders) | 10 (11) | 5 (10)
Salivary Hypersecretion (Gastrointestinal disorders) | 9 (10) | 3 (3)
Vomiting (Gastrointestinal disorders) | 14 (23) | 6 (8)
Blood Creatine Phosphokinase Increased (Investigations) | 8 (8) | 1 (1)
Akathisia (Nervous system disorders) | 27 (33) | 7 (7)
Headache (Nervous system disorders) | 8 (9) | 9 (13)
Tremor (Nervous system disorders) | 15 (18) | 4 (4)
Insomnia (Psychiatric disorders) | 20 (23) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No